CLINICAL TRIAL: NCT03391271
Title: The Use of Photobiomodulation Therapy for the Prevention of Chemotherapy-induced Peripheral Neuropathy: a Pilot Trial
Brief Title: PBMT for the Prevention of CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIPN-112017
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photobiomodulation therapy (PBMT) (Experimental): During photobiomodulation therapy (PBMT) or low-level laser therapy, visible and/or (near)-infrared laser light is used at the affected area to improve tissue repair and thereby promote functional recovery of peripheral nerves
  Interventions: Other: photobiomodulation therapy (PBMT)
- Placebo group (Placebo Comparator): No PBMT
  Interventions: Other: sham laser sessions

INTERVENTIONS:
Other: photobiomodulation therapy (PBMT) — Multiwave Locked System® (M6 laser, ASA srl, Arcugnano (VI), Italy)
  • The PBMT-group will receive twice-weekly laser sessions starting at first until the last week of chemotherapy (9-12 weeks depending on the type of chemotherapy)
  Arms: photobiomodulation therapy (PBMT)
Other: sham laser sessions — • The control group will undergo twice-weekly sham laser sessions starting at first until the last week of chemotherapy (9-12 weeks depending on the type of chemotherapy). The laser device will be placed on the same manner and for the same period of time on the identified body sites, but the device will not be switched on.
  Arms: Placebo group

SUMMARY:
ne of the most common cancers in women worldwide is breast cancer. A common used therapy in early-stage and metastatic breast cancer involves chemotherapy. Taxanes, microtubule-targeting agents (MTAs), are one of the most used chemotherapeutic agents in breast cancer patients. Unfortunately, this treatment comes with many unfortunate side effects. Chemotherapy-induced peripheral neuropathy (CIPN) is one of these common side effects. This condition involves paresthesia, numbness and/or burning pain in distal limbs. Eventually, loss of temperature sensation, loss of tendon reflexes and pain sensation can occur. Yet, no therapies have been developed to treat CIPN. At the moment, only symptom management is possible. Not only will this condition affect the patients' daily activities, but a chemotherapy dose reduction could also be necessary, influencing the outcome and overall survival rate of the patient.

A new and emerging treatment for CIPN is photobiomodulation therapy (PBMT) or low-level laser therapy. During PBMT, visible and/or (near)-infrared laser light is used at the affected area to improve tissue repair and thereby promote functional recovery of peripheral nerves. Studies have shown positive results for patients with diabetic neuropathy. However, no studies have been undertaken specifically for taxane-induced neuropathy (TIN).

We hypothesize that PBMT is an effective treatment strategy to prevent sensory symptoms associated with TIN. This can lead to an improved quality of life for the patient and no need for a chemotherapy dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-invasive (stage 0) or invasive (stage 1, 2 and 3A) breast adenocarcinoma
* Age 18 years or above
* Are planned to undergo at least 3 cycles of taxane treatment (i.e. paclitaxel or docetaxel)
* Have no documented or observable psychiatric or neurological disorders that might interfere with study participation (e.g., dementia or psychosis).
* Signed informed consent

Exclusion Criteria:

* Have a history of neuropathy before taxane treatment due to other medical conditions: diabetes, peripheral vascular disease, HIV infection, significant degenerative or familial neurologic disorder, nerve compression injuries (i.e., carpal tunnel syndrome, brachial plexopathy, spinal stenosis, or spinal nerve root compression)
* Taking stable doses of medication on prescription or dietary supplements for peripheral neuropathy. Related medications are: gabapentin, pregabalin, nortriptyline, amitriptyline, duloxetine, venlafaxine; lidocaine, opioid tramadol and other narcotics; NSAIDs; glutamine, glutathione, vitamin E and vitamin B12; Patients need to agree not to initiate a new therapy two weeks before and during the study period.
* Metastatic disease
* Have a diagnosis of ethanol addiction or dependence within the past 10 years.
* Concurrent chemotherapy with neurotoxic chemotherapeutic agents (i.e. platinum compounds or vinca alcaloids)
* Severe or unstable cardio- respiratory or musculoskeletal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
The modified total neuropathy score (mTNS) | baseline
  he mTNS is a composite scale that includes patient report of sensory and motor symptoms, pin sensibility, quantitative vibration thresholds, strength using manual muscle tests, and deep tendon reflexes. The higher the score, the more severe the peripheral neuropathy. The mTNS is a clinically applicable, sensitive screening tool for CIPN.
The modified total neuropathy score (mTNS) | week 6
  he mTNS is a composite scale that includes patient report of sensory and motor symptoms, pin sensibility, quantitative vibration thresholds, strength using manual muscle tests, and deep tendon reflexes. The higher the score, the more severe the peripheral neuropathy. The mTNS is a clinically applicable, sensitive screening tool for CIPN.
The modified total neuropathy score (mTNS) | week 12
  he mTNS is a composite scale that includes patient report of sensory and motor symptoms, pin sensibility, quantitative vibration thresholds, strength using manual muscle tests, and deep tendon reflexes. The higher the score, the more severe the peripheral neuropathy. The mTNS is a clinically applicable, sensitive screening tool for CIPN.
The modified total neuropathy score (mTNS) | week 15
  he mTNS is a composite scale that includes patient report of sensory and motor symptoms, pin sensibility, quantitative vibration thresholds, strength using manual muscle tests, and deep tendon reflexes. The higher the score, the more severe the peripheral neuropathy. The mTNS is a clinically applicable, sensitive screening tool for CIPN.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) | baseline
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) is a patient questionnaire to test the quality of life of the patients with taxane induced neuropathy (TIN) and can be divided into five components: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific for taxane treated patients. The higher the score, the better the quality of life.
Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) | week 6
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) is a patient questionnaire to test the quality of life of the patients with taxane induced neuropathy (TIN) and can be divided into five components: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific for taxane treated patients. The higher the score, the better the quality of life.
Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) | week 12
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) is a patient questionnaire to test the quality of life of the patients with taxane induced neuropathy (TIN) and can be divided into five components: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific for taxane treated patients. The higher the score, the better the quality of life.
Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) | week 15
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Taxane scale (FACT/GOG-Taxane) is a patient questionnaire to test the quality of life of the patients with taxane induced neuropathy (TIN) and can be divided into five components: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific for taxane treated patients. The higher the score, the better the quality of life.
Pain evaluation | baseline
  mechanical visual analogue scale (VAS) will be used to evaluate the patients' pain level due to TIN.
Pain evaluation | week 6
  mechanical visual analogue scale (VAS) will be used to evaluate the patients' pain level due to TIN.
Pain evaluation | week 12
  mechanical visual analogue scale (VAS) will be used to evaluate the patients' pain level due to TIN.
Pain evaluation | week 15
  mechanical visual analogue scale (VAS) will be used to evaluate the patients' pain level due to TIN.

CONTACTS AND LOCATIONS:
Overall Officials: jeroen Mebis, prof. dr., Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joy L, Jolien R, Marithe C, Stijn E, Laura S, Hilde L, Sandra B, Wendy N, Ruth H, Liesbeth R, Sylvana S, Sylvia H, Jeroen M. The use of photobiomodulation therapy for the prevention of chemotherapy-induced peripheral neuropathy: a randomized, placebo-controlled pilot trial (NEUROLASER trial). Support Care Cancer. 2022 Jun;30(6):5509-5517. doi: 10.1007/s00520-022-06975-x. Epub 2022 Mar 21. PMID 35312857